CLINICAL TRIAL: NCT01634360
Title: A 48-month Open Label Multi-centered Extension Study to Evaluate the Long-term Safety, Tolerability and Efficacy of E2007 in Patients With Parkinson's Disease With "Wearing Off" Motor Fluctuations and "on" Period Dyskinesias
Brief Title: Long-Term Safety, Tolerability and Efficacy in Perampanel Treated Parkinson's Disease Patients With Motor Fluctuations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to termination of clinical program for Parkinson's Disease
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-E044-205; 2004-000361-35 (EudraCT Number)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2013-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perampanel (1-4 mg) (Experimental): Subjects entered this open-label extension study from the double-blind core study (E2007-E044-204), and dosed placebo or perampanel. Subjects started this open-label extension study on perampanel 1 mg once daily for two weeks, followed by 2 mg once daily for two weeks; if they did not tolerate the 1 mg dose, subjects were withdrawn from the study. Subjects could be up-titrated to 3 or 4 mg in a sequential manner. Subjects could be down-titrated at any time to either 3, 2 or 1 mg in a sequential manner.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — 1mg once daily for two weeks, followed by 2mg once daily for 2 weeks; if they did not tolerate the 1 mg dose, subjects were withdrawn from the study. Subjects could be up-titrated to 3 or 4 mg in a sequential manner. Subjects could be down-titrated at any time to either 3, 2 or 1 mg in a sequential manner.
  Other Names: E2007

SUMMARY:
A 48-month open label multi-centered extension study to evaluate the long-term safety, tolerability and efficacy of E2007 in patients with Parkinson's Disease with "wearing off" motor fluctuations and "on" period Dyskinesias.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in Study E2007-E044-204 and who either completed 12 weeks of study drug treatment or who withdrew from the study due to lack of efficacy.

Exclusion Criteria:

* Pregnant or lactating women.
* Women of child bearing potential unless infertile (including surgically sterile) or practicing effective contraception (e.g. abstinence, IUD-intrauterine device, or barrier method plus hormonal method). These patients must also be willing to remain on their current form of contraception for the duration of the study. Postmenopausal women may be recruited but must be amenorrhoeic for at least 1 year to be considered of non-child bearing potential.
* Fertile men not willing to use reliable contraception and fertile men with partners not willing to use reliable contraception. These patients and their partners must also be willing to remain using reliable contraception for the duration of the study.
* Patients with a past or present history of drug or alcohol abuse.
* Patients with a past (within one year) or present history of psychotic symptoms requiring antipsychotic treatment. Patients may be taking anti-depressant medication, however the dose must have been kept stable for at least 8 weeks prior to baseline visit.
* Patients with unstable abnormalities of the hepatic, renal, cardiovascular, respiratory, gastro-intestinal, haematological, endocrine or metabolic systems which might complicate assessment of the tolerability of the study medication.
* Patients with significantly elevated liver enzymes (abnormal bilirubin or serum transaminase levels of more than 1.5 times the upper normal limit).
* Patients with current or prior treatment (within 4 weeks prior to the Baseline visit) with medication known to induce the enzyme cytochrome P450 3A4 including but not limited to; carbamazepine; dexamethasone; ethosuximide; phenobarbital; phenytoin; primidone; rifabutin; rifampicin; and St John's Wort.
* Current or prior treatment (within 4 weeks prior to baseline visit) with methyldopa, budipine, reserpine or intermittent use of liquid forms of levodopa or as needed (prn) apo-morphine.
* Patients with previous stereotactic surgery (e.g. pallidotomy) for Parkinson's disease or who are likely to undergo surgery for Parkinson's disease while participating in this study.
* Patients receiving deep brain stimulation (DBS) or who are likely to undergo DBS for Parkinson's disease while participating in the extension study.
* Patients with clinically significant cognitive impairment (mini-mental state examination (MMSE) <24 and /or fulfilling diagnostic and statistical manual of mental disorders (DSM IV) criteria for dementia due to Parkinson's disease).
* Patients with conditions affecting the peripheral or central sensory system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel (Placebo During Core Study); Perampanel (Perampanel 0.5, 1, or 2 mg During Core Study): Subjects entered this open-label extension study from the double-blind core study (E2007-E044-204). Subjects started on perampanel 1mg once daily for 4 weeks, followed by 2mg once daily for 2 weeks; if they did not tolerate the 1 mg dose, subjects were withdrawn from the study. Subjects could be up-titrated to 3 or 4 mg in a sequential manner. There were at least 2 weeks between each titration to assess safety and tolerability, and the subjects attended a clinic visit for safety review and dispensing of more medication. Subjects could be down-titrated at any time to either 3, 2 or 1 mg in a sequential manner.
Period: Overall Study
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 0.5, 1, or 2 mg During Core Study)
Started | 49 | 136
Completed | 0 | 0
Not Completed | 49 | 136
Not completed — Adverse Event | 10 | 34
Not completed — subject withdrew consent | 13 | 23
Not completed — Protocol Violation | 1 | 1
Not completed — Lack of Efficacy | 4 | 14
Not completed — Other | 3 | 20
Not completed — Study termination by sponsor | 18 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 0.5, 1, or 2 mg During Core Study) | Total
Number analyzed (Participants) | 48 | 134 | 182
Age, Customized [Number; unit: Participants] — Safety population
  Participants
    <65 years | 27 | 72 | 99
    >=65 years | 21 | 62 | 83
Sex: Female, Male [Count of Participants; unit: Participants] — The participant flow information was collected from all participants who entered the study. Baseline information was collected only for the safety population (all subjects who received at least 1 dose of perampanel in this study and at least 1 dose of study medication during the double-blind phase of the core study).
  Participants
    Female | 23 | 54 | 77
    Male | 25 | 80 | 105
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    Caucasian | 48 | 134 | 182

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Daily OFF Time (Hours) During Open-label Extension Study
Description: OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor. This outcome measure was based on data collected through use of a patient diary.
Time Frame: Baseline, Week 0, Week 12, Week 24, Week 36, Week 52, Week 78, Week 104, Week 130, Week 156
Population: Efficacy Population- All subjects who were in the Safety Population and for whom at least 1 postbaseline (post Week 0) efficacy assessment was made.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 0.5, 1, or 2 mg During Core Study)
Number analyzed (Participants) | 45 | 125
Hours
  Week 0 | -0.51 (2.811) | -0.68 (2.479)
  Week 12 | -0.91 (2.913) | -1.08 (2.907)
  Week 24 | -1.05 (2.760) | -1.15 (2.754)
  Week 36 | -0.76 (2.638) | -1.16 (2.959)
  Week 52 | -0.47 (3.443) | -1.34 (2.881)
  Week 78 | -1.31 (2.547) | -1.54 (3.106)
  Week 104 | -1.14 (3.121) | -1.81 (3.149)
  Week 130 | -0.65 (3.710) | -1.62 (2.953)
  Week 156 | -1.00 (2.953) | -1.16 (2.672)

2. Secondary Outcome: Mean Change From Baseline in Total Daily ON Time (Without Dyskinesias or With Non-troublesome Dyskinesias) (Hours) During Open-label Extension Study
Description: ON state is when medication is providing benefits with regard to stiffness, slowness, and tremor. This outcome measure was based on data collected through use of a patient diary.
Time Frame: Baseline, Week 0, Week 12, Week 24, Week 36, Week 52, Week 78, Week 104, Week 130, Week 156
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 0.5, 1, or 2 mg During Core Study)
Number analyzed (Participants) | 45 | 125
Hours
  Week 0 | 0.85 (2.856) | 1.17 (3.562)
  Week 12 | 1.47 (3.200) | 1.32 (3.758)
  Week 24 | 1.89 (3.712) | 0.86 (3.632)
  Week 36 | 1.40 (3.895) | 1.52 (4.153)
  Week 52 | 0.81 (4.101) | 1.79 (4.238)
  Week 78 | 1.39 (4.450) | 2.52 (4.625)
  Week 104 | 0.21 (4.541) | 3.30 (4.617)
  Week 130 | -0.98 (4.276) | 1.42 (4.013)
  Week 156 | -0.73 (4.105) | 1.76 (4.974)

3. Secondary Outcome: Mean Change From Baseline in UPDRS Part III (Motor) Score in ON State (Hours) During Open- Label Extension Study
Description: Unified Parkinson's Disease Rating Scale (UPDRS) is a standardized assessment of the symptoms and signs of Parkinson's Disease. Part III assesses motor activity, based on 14 items, such as gait, facial expression, and rigidity. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms. Range of possible total scores, 0 to 56.
  ON state is when medication is providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline, Week 0, Week 12, Week 24, Week 36, Week 52, Week 78, Week 104, Week 130, Week 156
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 0.5, 1, or 2 mg During Core Study)
Number analyzed (Participants) | 45 | 125
Scores on scale
  Week 0 | 2.30 (6.360) | 1.46 (7.501)
  Week 12 | 2.45 (6.926) | 0.36 (7.137)
  Week 24 | 2.43 (7.247) | 1.80 (7.912)
  Week 36 | 2.69 (8.177) | 2.78 (9.602)
  Week 52 | 2.76 (6.947) | 3.83 (9.084)
  Week 78 | 3.64 (7.279) | 3.43 (9.344)
  Week 104 | 6.25 (9.345) | 4.11 (10.999)
  Week 130 | 6.05 (9.610) | 2.77 (9.680)
  Week 156 | 5.72 (8.115) | 4.20 (9.034)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAE) are those that start on or after the first day of dosing with study medication in the open label extension study, and no later than 30 days after the last day of dosing with study medication.
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 0.5, 1, or 2 mg During Core Study)
Serious Adverse Events (participants affected / at risk) | 13/48 | 39/134
Other Adverse Events (participants affected / at risk) | 3/48 | 0/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (Placebo During Core Study) (N=48) | Perampanel (Perampanel 0.5, 1, or 2 mg During Core Study) (N=134)
Dyskinesia (Nervous system disorders) | 0 | 3
On and off phenomenon (Nervous system disorders) | 1 | 2
Dementia (Nervous system disorders) | 0 | 2
Balance disorder (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dystonia (Nervous system disorders) | 1 | 0
Freezing phenomenon (Nervous system disorders) | 0 | 1
Hyperkinesia (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0
Psycomotor hyperactivity (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Posture abnormal (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 3
Confusional state (Psychiatric disorders) | 0 | 2
Hallucination, visual (Psychiatric disorders) | 1 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 1 | 0
Dissociation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Device malfunction (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerous fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Radial nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Benign ovarian tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostrate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Arterial stenosis limb (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1
Blood alkaline phosphatase (Investigations) | 0 | 1
Blood pressure decrease (Investigations) | 1 | 0
Heamatocrit decreased (Investigations) | 0 | 1
Investigation (Investigations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Social stay hospitalisation (Social circumstances) | 1 | 1
Deep brain stimulation (Surgical and medical procedures) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (Placebo During Core Study) (N=48) | Perampanel (Perampanel 0.5, 1, or 2 mg During Core Study) (N=134)
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Due to early termination, no subjects completed this open-label extension study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No